CLINICAL TRIAL: NCT01539005
Title: Is Tuberculosis Recurrence in Treated Tuberculosis-Human Immunodeficiency Virus (HIV) Co-Infected Patients Relapse or Re-infection?
Brief Title: Tuberculosis Recurrence Upon Treatment With Highly Active Antiretroviral Therapy
Acronym: TRuTH
Status: Completed | Type: Observational
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency); Howard Hughes Medical Institute (Other); K-RITH (Other)
Responsible Party: Principal Investigator, Dr Kogieleum Naidoo, Principal Investigator, Centre for the AIDS Programme of Research in South Africa
Other Study IDs: CAP005
Record Dates: First submitted 2012-02-10; First posted 2012-02-27 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Tuberculosis
Keywords: Recurrence; Tuberculosis
MeSH Terms: conditions — Tuberculosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored Plasma/Serum/PBMCs: Participants who consent to have additional samples stored for future testing will have serum, plasma and PBMCs stored . Possible uses of plasma include assessment of host genetics profiles, including HLA profile, additional viral load assays.Possible uses of serum include additional safety serology and evaluation of suspected IRIS on participants where indicated. The PBMCs will be used to test for IRIS/PR when suspected.
  Other potential tests that may be performed on the stored specimens include new generation assays of immunity.
  Stored Sputum Isolates :RFLP testing will be performed from stored bacterial isolates on all positive cultures in which recurrence is suspected and compared to the initial positive culture used to diagnose the TB initially.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a cohort observational study investigating the rate of tuberculosis (TB) recurrence in adult patients who have completed TB therapy for Pulmonary TB (PTB) and are on highly active antiretroviral therapy (HAART).The primary objective of this study is to determine the incidence of TB recurrence in patients on HAART.The study is being conducted at the CAPRISA eThekwini Clinical Research Site (CRS), which is adjacent to the Prince Cyril Zulu Communicable Disease Clinic (PCZCDC), a major urban TB clinic, in Durban, South Africa.No hypotheses will be tested in this study; however, the primary study question will determine the proportion of TB recurrence due to relapse vs. re-infection.The study has enrolled 402 participants

DETAILED DESCRIPTION:
1. Objective: To determine the extent of and reasons for relapse and re-infection in incident cases of tuberculosis (TB) in Human Immunodeficiency Virus (HIV)-infected patients on Highly Active Antiretroviral Therapy (HAART)
2. Design: A prospective cohort study of patients with HIV previously treated for pulmonary TB and initiated on HAART in the SAPIT (Starting AIDS treatment at three Points in TB treatment) and START (Starting Tuberculosis and Anti-Retroviral Therapy) trials. Each incident case of TB recurrence in this cohort of adult patients on HAART will be investigated to assess whether the infecting mycobacterium is similar to that from the previous infection and whether the immune responses differ in cases of relapse and re-infection.
3. Population: Men and women 18 years of age with documented HIV infection and past TB therapy as part of the SAPIT and START trial will be enrolled.
4. Study Procedures: This study will involve 3 years of follow-up of patients who had been initiated on a course of TB therapy as part of the SAPIT and START trials. Upon exit from the SAPIT trial (i.e. 18 months post-TB diagnosis), study patients will be consented and enrolled in this cohort study. Study participants will be seen monthly for the first 3 months and thereafter 3 monthly, for routine clinic visits and ART services. At every visit patients will be screened for TB recurrence clinically, with chest radiograph and, whenever possible, with available TB diagnostics or new diagnostics that are being developed and/or tested.
5. Study Outcome The primary endpoint of this study will be the development of recurrent TB. TB recurrence as a result of relapse will be defined as isolates of M. tuberculosis from the first and second episodes of TB which cluster in Restriction Fragment Length Polymerization (RFLP) analysis. TB recurrence as a result of re-infection will be defined as isolates from the first and second episode of TB which differ on RFLP analysis. Each study participant who has recurrent TB will be assessed by Interferon (IFN) gamma ELISPOT assay to compare cytotoxic lymphocyte (CTL)immune responses in TB relapse and re-infection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (> 18 years) who were diagnosed as co-infected with TB and HIV and previously enrolled in the SAPIT and START trials
2. Willing to consent to participate in this study and contribute specimens to the K-RITH repository for future investigations

Exclusion Criteria:

1. Patients with Extensively drug-resistant (XDR) TB will not be eligible.
2. Patients who refuse consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women > 18 years of age with documented HIV infection and past TB therapy as part of the SAPIT and START trial will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2009-11; Primary Completion 2014-04-23 (Actual); Study Completion 2014-04-23 (Actual)

PRIMARY OUTCOMES:
Tuberculosis | Tuberculosis case finding will be conducted over a 36 month period. Tuberculosis investigations will be conducted from the date of Enrollment to the date of TB diagnosis based on a positive sputum TB culture
  The primary endpoint of this study will be development of TB. TB recurrence as a result of relapse will be defined as isolates of M.tuberculosis from the first and second episodes of TB which cluster in Restriction Fragment Length Polymerization analysis. TB recurrence as a result of re-infection will be defined as isolates from the first and second episode of TB which differ on RFLP analysis. To detect TB, patients will have a sputum smear at every study visit. Chest X-Ray and safety bloods are conducted 6-monthly.

CONTACTS AND LOCATIONS:
Overall Officials: Kogieleum Naidoo, MBChB, Principal Investigator — Centre for the AIDS Programme of Research in South Africa; Salim S Abdool Karim, MBChB, PhD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- CAPRISA eThekwini Clinical Research Site, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Fischinger S, Cizmeci D, Shin S, Davies L, Grace PS, Sivro A, Yende-Zuma N, Streeck H, Fortune SM, Lauffenburger DA, Naidoo K, Alter G. A Mycobacterium tuberculosis Specific IgG3 Signature of Recurrent Tuberculosis. Front Immunol. 2021 Sep 22;12:729186. doi: 10.3389/fimmu.2021.729186. eCollection 2021. PMID 34630406